CLINICAL TRIAL: NCT00942396
Title: Study to Compare the Diagnostic Accuracy of Nuance Full-Field Digital Mammography to Screen-Film Mammography
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA changed classification of device and no longer requires this type of clinical data
Sponsor: Planmed Oy (Industry)
Responsible Party: Chris Oldham/ Director of North American Sales, Planmed OY
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TK01007
Record Dates: First submitted 2009-07-07; First posted 2009-07-20 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Breast Cancer
Keywords: Mammography
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mammography (Experimental): Women must be at least 40 years of age, presenting for routine breast cancer screening or presenting with one or both breasts scored 4 or 5 on the BI-RADS scale as a result of SFM either for routine breast cancer screening or for follow-up or diagnostic mammography
  Interventions: Device: Full Field Digital Mammogram (Planmed Sophie Nuance)

INTERVENTIONS:
Device: Full Field Digital Mammogram (Planmed Sophie Nuance) — Full Field Digital Mammogram
  Other Names: mammography; digital mammography

SUMMARY:
Evaluate the diagnostic accuracy of the Planmed Sophie Nuance Full Field Digital Mammography (FFDM) X-ray System compared to screen-film mammography (SFM) in the detection of breast cancer.

DETAILED DESCRIPTION:
Objectives: 1) To establish the non-inferiority of the diagnostic accuracy of the Planmed Sophie Nuance Full Field Digital Mammography (FFDM) X-ray System compared to screen-film mammography (SFM) in the detection of breast cancer; and 2) To demonstrate in a comparative side-by-side feature analysis that interpretations based on the Planmed Sophie Nuance FFDM X-ray System are diagnostically non-inferior to SFM in the detection of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 40 years of age or older
2. Subject is presenting for routine breasts cancer screening (Cohort I) OR Subject has one or both breasts scored 4 or 5 on the BI-RADS scale as a result of SFM either for routine breast cancer screening or for follow-up or diagnostic mammography (Cohort II)
3. Subject's schedule permits the SFM and the FFDM to be performed no more than 30 days apart and with no intervention between the exams
4. Subject will provide prospective, written informed consent
5. Subject is considered capable of complying with study procedures including a willingness to return for a one-year follow-up exam -

Exclusion Criteria:

1. Subject is pregnant or possibly pregnant or planning pregnancy within the next 15 months
2. Subject has undergone a breast augmentation or breast implant? Has subject had any of the following breast procedures?

   Fine needle or cyst aspiration NOT Eligible if within past year Biopsy Not Eligible if within past year Lumpectomy (for breast cancer) Mastectomy (for breast cancer) Radiation therapy Breast reconstruction Breast reduction Not Eligible if within past year
3. Subject has had an invasive breast procedure or operation within the past year
4. Subject has significant existing breast trauma
5. Subject has a history of breast cancer treated with operation or radiation
6. Subject has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete good quality data

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Area under ROC curve based on subjects' maximum POM scores; sensitivity based on subjects' maximum BI-RADS scores with 4 or higher as positive for cancer; and specificity based on subjects maximum BI-RADS scores with 4 or higher as positive for cancer | Approximately one year after completion of study.

SECONDARY OUTCOMES:
area under the ROC curve based on the maximum POM score per subject-breast | Approximately one year after completion of study.
area under the ROC curve based on the POM scores from the ten regions of a subject's breasts; | Approximately one year after completion of study.
sensitivity based on subjects' maximum BI-RADS scores using a cut-point of 3 or higher as positive for cancer; | Approximately one year after completion of study.
specificity based on subjects' maximum BI-RADS scores using a cut-point of 3 or higher as positive for cancer; | Approximately one year after completion of study.
Sensitivity and specificity based on the maximum BI-RADS scores per subject-breast using 4 or higher for positive; and sensitivity and specificity based on the maximum BI-RADS scores per subject-breast using 3 or higher for positive. | Approximately one year after completion of study.
Feature Analysis Study; side by side assessment of SFM and FFDM images and comparison of quality features: lesion conspicuity, tissue visibility at chest wall, tissue visibility at skin line, axillary details (MLO), overall contrast, overall sharpness | Approximately one year after completion of study.
Adverse event assessment | Approximately 24 hours after completion of FFDM

CONTACTS AND LOCATIONS:
Overall Officials: Sami Tohka, PhD, Study Director — Planmed Oy
Locations (2):
- United States (2):
  - Mroz-Baier Breast Care Clinic, Memphis, Tennessee
  - The Rose, Houston, Texas